CLINICAL TRIAL: NCT00313183
Title: A Randomized, Single-Blind, Dose-Rising, Placebo-Controlled, Crossover Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of SYMLIN in Adolescent Subjects With Type 1 Diabetes Mellitus
Brief Title: A Study to Evaluate Symlin in Adolescent Subjects With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 137-162
Record Dates: First submitted 2006-04-10; First posted 2006-04-12 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-01

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes; pediatric; pramlintide; Symlin; Amylin
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — pramlintide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): single doses of pramlintide acetate or placebo, given in three different sequences to three cohorts of subjects
  Interventions: Drug: pramlintide acetate

INTERVENTIONS:
Drug: pramlintide acetate — single subcutaneous doses of 15mcg and 30mcg
  Other Names: Symlin

SUMMARY:
This study will be the first evaluation of Symlin in adolescent subjects with type 1 diabetes mellitus and is designed to evaluate the blood levels (pharmacokinetics), biochemical and physiological effects (pharmacodynamics), and safety and tolerability of Symlin in these subjects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 1 diabetes mellitus for at least 1 year prior to screening
* Be on a stable regimen requiring multiple daily injections of basal and mealtime insulin or continuous subcutaneous insulin infusion for at least 2 weeks prior to screening
* HbA1c between 6.0% and 10.0%, inclusive, at screening
* Body weight >=50 kg at screening

Exclusion Criteria:

* Currently being treated with the following medications: *Any oral antihyperglycemic agent; *Drugs that directly affect gastrointestinal motility
* Has been previously treated with Symlin/pramlintide (or has participated in a Symlin/pramlintide clinical study)
* Has received any investigational drug within 1 month of screening

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2006-04; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the pharmacokinetics of Symlin in adolescent subjects with type 1 diabetes | single doses
To assess the safety and tolerability of Symlin in adolescent subjects with type 1 diabetes | single doses

SECONDARY OUTCOMES:
To evaluate the effects of Symlin compared to placebo in adolescent subjects with type 1 diabetes on various pharmacodynamic endpoints | single doses

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Porter, MD, Study Director — Amylin Pharmaceuticals, LLC.
Locations (3):
- United States (3):
  - Research Site, Aurora, Colorado
  - Research Site, Kansas City, Missouri
  - Research Site, New York, New York